CLINICAL TRIAL: NCT02229305
Title: Child System and Treatment Enhancement Projects (Child STEPs); The Clinic Treatment Project in Maine - Phase III
Brief Title: Maine Implementation Study - Phase III
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard University (Other)
Collaborators: MacArthur Foundation (Other); Casey Family Programs (Unknown); Annie E. Casey Foundation (Other Government)
Responsible Party: Principal Investigator, John Weisz, Primary Investigator, Harvard University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STEPs Phase III
Record Dates: First submitted 2014-08-28; First posted 2014-09-01 (Estimated); Last update posted 2014-09-01 (Estimated); Status verified 2014-08

CONDITIONS: Anxiety; Trauma; Depression; Problem Behavior
Keywords: Anxiety; Trauma; Depression; Problem Behavior; evidence-based treatments
MeSH Terms: conditions — Anxiety Disorders; Wounds and Injuries; Depression; Problem Behavior

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual Care Treatment (Active Comparator): Usual Care therapists could use any treatment procedures they used regularly in their clinical practice.
  Interventions: Behavioral: Usual Care Treatment
- Modular Approach to Therapy for Children (Experimental): Therapists used a modular manual (Modular Approach to Therapy for Children with Anxiety, Depression, Trauma, or Conduct Problems; Chorpita & Weisz, 2010) to help children with primary problems of anxiety, depression, trauma, and conduct.
  Interventions: Behavioral: Modular Approach to Therapy for Children

INTERVENTIONS:
Behavioral: Usual Care Treatment — Usual Care therapists could use any treatment procedures they used regularly in their clinical practice.
  Arms: Usual Care Treatment
Behavioral: Modular Approach to Therapy for Children — Therapists used the Modular Approach to Therapy for Children with Anxiety, Depression, Trauma, or Conduct Problems (MATCH-ADTC; Chorpita & Weisz, 2010).
  Arms: Modular Approach to Therapy for Children

SUMMARY:
This study focused on youths who were referred to community-based mental healths clinics for problems related to disruptive behaviors, depression, anxiety, traumatic stress, and any combination of these problems. Therapists were randomly assigned to deliver usual treatment procedures (usual care, or UC) in their clinics or an evidence-based, modularized treatment (Modular Approach to Therapy for Children with Anxiety, Depression, Trauma, or Conduct Problems, or MATCH-ADTC). Assessments were conducted at pre-treatment and post-treatment, and every 3 to 6 months for two years. Results will address critical questions about deployment of evidence-based youth practices to clinical settings.

DETAILED DESCRIPTION:
This study focused on youths aged 6 - 15 who were referred to community-based mental healths clinics for problems related to disruptive behaviors, depression, anxiety, traumatic stress, and any combination of these problems. Using a randomized block design, therapists were randomly assigned to deliver usual treatment procedures (usual care, or UC) in their clinics or an evidence-based, modularized treatment (Modular Approach to Therapy for Children with Anxiety, Depression, Trauma, or Conduct Problems, or MATCH-ADTC). MATCH-ADTC was supported by training and supervision procedures designed to fit providers and their clinic contexts. Assessments were carried out at pre-treatment, at post-treatment, and at 3-,6-,9-,12,18-,and 24-month follow-ups. Assessments carried out at pre-treatment included (a) individual youth problems and disorders; (b) individual youth functioning at home and school; and (c) clinic staff beliefs and attitudes toward evidence-based treatments. Assessments carried out at post-treatment and follow-ups included measures of (1) youth, caregiver, and therapist satisfaction with treatment; (b) youth, caregiver, and therapist views on the quality of the therapeutic relationship; and (c) treatment costs. Assessments carried out at follow-up only included measures of (a) caregiver reports of any mental health service use following project treatment; (b) therapist reports on the extent to which the treatment procedures they used in the project are continued after project termination. Analyses will address critical questions about deployment of evidence-based youth practices to clinical settings.

ELIGIBILITY:
Inclusion Criteria:

* 6 - 15 year old and their caregivers
* seeking services at community mental health clinics
* primary problem or disorder related to anxiety, traumatic stress, depression, or conduct problems, or any combination of the four problems

Exclusion Criteria:

* Child is younger than 6 years or older than 15 years on the day of the phone screen
* Child has attempted suicide within the past year
* Schizophrenic spectrum disorders (including MDD with psychotic features)
* Autism or another Pervasive Developmental Disorder (E.g., PDD NOS, Asperger's Disorder, Child Disintegration Disorder, Rett's Disorder)
* Anorexia Nervosa
* Bulimia Nervosa
* Mental Retardation
* No relevant T-scores validate target disorders
* ADHD identified as primary reason for seeking treatment at phone screen
* Child's medication has not been regulated for one month or longer

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 235 (Actual)
Dates: Start 2008-12; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Brief Problem Checklist (BPC, parent and child forms) | Change over time from Day 1 to Day 242 (end of treatment)
  Youth and parents were contacted weekly to report changes in youth functioning. Each person was asked to rate their own or their child's behavior on 12 items (6 internalizing and 6 externalizing behaviors) that were adapted from the Youth Self Report and the Child Behavior Checklist. Children and caregivers completed the pre-treatment assessment on Day 1, every week during treatment, and at post-treatment assessment which occurred on average 242days (SD = 121 days) after the pre-treatment assessment.
Top Problems Assessment | Change over time from Day 1 to Day 735 (24-month follow-up)
  Youths and parents were asked to identify "The three most important problems for which you need [or "your child needs"] help." at the intake assessment. The six resulting problems (3 from youth, 3 from parent) were then rated on a scale of 0 ("Not serious at all") to 10 ("Very serious problem") by youth and parent. Youths and parents completed the pre-treatment assessment on Day 1, at post-treatment assessment which occurred on average 242 days (SD = 121 days) after the pre-treatment assessment, and at 3-, 6-, 9-, 12- and 24-month follow-up from Day 1. (Used as a measure of clinical outcome.)

SECONDARY OUTCOMES:
UCLA PTSD Index | Change over time from Day 1 to Day 735 (24-month follow-up)
  The PTSD Index is a 38-item questionnaire that is widely-used to assess post-traumatic stress symptoms in children. Part I is a brief lifetime trauma screen. If a significant trauma is identified, Part II assesses DSM-IV PTSD symptoms related to the trauma. Part III assesses frequency of post-traumatic stress symptoms during the past month. The measure has shown good convergent validity, strong test-retest reliability, and Cronbach's alpha values in the .90s. We will administer it separately to students and their caregivers at pre-treatment, to determine whether post-traumatic stress should be a focus of treatment, and we will re-administer it at post-treatment and follow-up to assess change over time. Youths and parents completed the pre-treatment assessment on Day 1, at post-treatment assessment which occurred on average 242 days (SD = 121 days) after the pre-treatment assessment, and at 3-, 6-, 9-, 12- and 24-month follow-up from Day 1. (Used as a measure of clinical outcome.)
Youth Self Report (YSR) | Change over time from Day 1 to Day 735 (24-month follow-up)
  The YSR assesses problems in children on eight narrow-band scales (Withdrawn, Somatic Complaints, Anxious, Social Problems, Thought Problems, Attention Problems, Rule-Breaking Behavior, Aggressive Behavior), three broad-band scales (Internalizing, Externalizing, and Total problems), and six DSM-oriented scales. Children completed the pre-treatment assessment on Day 1, at post-treatment assessment which occurred on average 242 days (SD = 121 days) after the pre-treatment assessment, and at 3-, 6-, 9-, 12- and 24-month follow-up from Day 1.(Used as a measure of clinical outcome.)
Child Behavior Checklist | Change over time from Day 1 to Day 735 (24-month follow-up)
  The CBCL assesses problems in children on eight narrow-band scales (Withdrawn, Somatic Complaints, Anxious, Social Problems, Thought Problems, Attention Problems, Rule-Breaking Behavior, Aggression), three broad-band scales (Internalizing, Externalizing, and Total problems), and six DSM-oriented scales. Caregivers completed the pre-treatment assessment on Day 1, at post-treatment assessment which occurred on average 267 days (SD = 124 days) after the pre-treatment assessment, and at 3-, 6-, 9-, 12- and 24-month follow-up from Day 1. (Used as a measure of clinical outcome.)
Therapeutic Alliance Scale for Children | Post-treatment (Day 267)
  The quality of youths' working alliance with their therapists was assessed via the Therapeutic Alliance Scale for Children (TASC, Shirk & Saiz, 1992). The 7-item scale comes in both a youth-report form and a parent-report form (parents reporting on their youth's relationship with the therapist). On average, children and caregivers completed the post-treatment assessment 267 days (SD = 124 days) after the pre-treatment assessment. (Available for supplemental analyses.)
Service Assessment for Children and Adolescents: Treatment and Auxiliary Service Use Scales | Change over tiem from Day 1 to Day 735 (24-month follow-up)
  The SACA (Horwitz et al., 2001)is a standardized interview for youths and parents that measures use of mental health services across a broad spectrum (including outpatient, inpatient, and school-based). SACA reliability and validity data are well-documented. Caregivers completed the pre-treatment assessment on Day 1, at post-treatment assessment which occurred on average 267 days (SD = 124 days) after the pre-treatment assessment, and at 12- and 24-month follow-up from Day 1.(Available for supplemental analyses.)
Brief Impairment Scale | Change over time from Day 1 to Day 735 (24-month follow-up)
  The BIS is a 23-item instrument that evaluates three domains of functioning: interpersonal relations, school/work functioning, and self-care/self-fulfillment. Its advantages over other global impairment instruments are that it is respondent based, short in administration time, and multidimensional. Caregivers completed the pre-treatment assessment on Day 1, at post-treatment assessment which occurred on average 267 days (SD = 124 days) after the pre-treatment assessment, and at 12- and 24-month follow-up from Day 1.(Available for supplemental analyses.)
Services for Children and Adolescents - Parent Interview (SCAPI) | Change over time from Day 1 to Day 735 (24-month follow-up)
  The SCAPI is a measure that tracks child's use of medication as reported by the parent. Caregivers completed the pre-treatment assessment on Day 1, at post-treatment assessment which occurred on average 267 days (SD = 124 days) after the pre-treatment assessment, and at 3-, 6-, 9-, 12- and 24-month follow-up from Day 1.(Available for supplemental analyses.)

CONTACTS AND LOCATIONS:
Overall Officials: John R Weisz, PhD, Principal Investigator — Harvard University
Locations (1):
- Judge Baker Children's Center, Boston, Massachusetts, United States

REFERENCES:
- [Background] Chorpita BF, Bernstein A, Daleiden EL; Research Network on Youth Mental Health. Driving with roadmaps and dashboards: using information resources to structure the decision models in service organizations. Adm Policy Ment Health. 2008 Mar;35(1-2):114-23. doi: 10.1007/s10488-007-0151-x. Epub 2007 Nov 6. PMID 17987376
- [Background] Borntrager CF, Chorpita BF, Higa-McMillan C, Weisz JR. Provider attitudes toward evidence-based practices: are the concerns with the evidence or with the manuals? Psychiatr Serv. 2009 May;60(5):677-81. doi: 10.1176/ps.2009.60.5.677. PMID 19411357
- [Background] Ebesutani C, Bernstein A, Nakamura BJ, Chorpita BF, Higa-McMillan CK, Weisz JR; The Research Network on Youth Mental Health. Concurrent Validity of the Child Behavior Checklist DSM-Oriented Scales: Correspondence with DSM Diagnoses and Comparison to Syndrome Scales. J Psychopathol Behav Assess. 2010 Sep;32(3):373-384. doi: 10.1007/s10862-009-9174-9. Epub 2009 Nov 27. PMID 20700377
- [Background] Chorpita BF, Reise S, Weisz JR, Grubbs K, Becker KD, Krull JL; Research Network on Youth Mental Health. Evaluation of the Brief Problem Checklist: child and caregiver interviews to measure clinical progress. J Consult Clin Psychol. 2010 Aug;78(4):526-36. doi: 10.1037/a0019602. PMID 20658809
- [Background] Ebesutani C, Chorpita BF, Higa-McMillan CK, Nakamura BJ, Regan J, Lynch RE. A psychometric analysis of the Revised Child Anxiety and Depression Scales--parent version in a school sample. J Abnorm Child Psychol. 2011 Feb;39(2):173-85. doi: 10.1007/s10802-010-9460-8. PMID 20878460
- [Background] Palinkas LA, Schoenwald SK, Hoagwood K, Landsverk J, Chorpita BF, Weisz JR; Research Network on Youth Mental Health. An ethnographic study of implementation of evidence-based treatments in child mental health: first steps. Psychiatr Serv. 2008 Jul;59(7):738-46. doi: 10.1176/ps.2008.59.7.738. PMID 18586990
- [Background] Weisz JR, Chorpita BF, Palinkas LA, Schoenwald SK, Miranda J, Bearman SK, Daleiden EL, Ugueto AM, Ho A, Martin J, Gray J, Alleyne A, Langer DA, Southam-Gerow MA, Gibbons RD; Research Network on Youth Mental Health. Testing standard and modular designs for psychotherapy treating depression, anxiety, and conduct problems in youth: a randomized effectiveness trial. Arch Gen Psychiatry. 2012 Mar;69(3):274-82. doi: 10.1001/archgenpsychiatry.2011.147. Epub 2011 Nov 7. PMID 22065252
- See also: Child System and Treatment Enhancement Projects — http://www.child-steps.org/